CLINICAL TRIAL: NCT06359002
Title: A First-in-human Dose Escalation and Expansion Trial With the Antibody-drug Conjugate BYON4413 to Evaluate Safety, Pharmacokinetics, and Preliminary Efficacy in Patients With Relapsed/Refractory Acute Myeloid Leukemia or Myelodysplastic Neoplasms.
Brief Title: Safety, Pharmacokinetics, and Preliminary Efficacy of BYON4413 in Acute Myeloid Leukemia and Myelodysplastic Neoplasms.
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Byondis B.V. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BYON4413.001; 2023-507781-13-00 (EU CTIS Number)
Record Dates: First submitted 2024-03-26; First posted 2024-04-11 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Relapsed / Refractory AML; Relapsed / Refractory MDS
Keywords: BYON4413; CD123; Hematologic Malignancies; Antibody Drug Conjugate; AML; MDS
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence; Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose Escalation (Experimental): Escalating dose cohorts of BYON4413 for patients with AML or MDS.
  Interventions: Drug: BYON4413

INTERVENTIONS:
Drug: BYON4413 — BYON4413 will be administered by IV infusion.

SUMMARY:
This is the first-in-human trial with BYON4413 to evaluate safety, PK, immunogenicity, and anti-leukemia activity of BYON4413 in patients with AML or MDS.

DETAILED DESCRIPTION:
This trial includes two parts. Part 1 is a dose escalation study in which the maximum tolerated dose and recommended dose for expansion of BYON4413 will be determined. Part 2 is an expansion study to evaluate the anti-leukemia activity and safety of BYON4413.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have progressed on standard therapy or have no established alternative treatment, with a diagnosis of:

  * R/R AML (WHO 2022) OR
  * MDS (WHO 2022) with ≥10% blasts in BM and have received ≥3 cycles of HMA
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2;
* Adequate baseline organ function.

Exclusion Criteria:

* Having been treated with any CD123-targeting therapies;
* Having received allogeneic hematopoietic stem cell transplantation within 100 days prior to start Cycle 1 Day 1;
* Having treatment-related toxicities from prior anti-leukemia therapies that have not resolved to CTCAE Grade ≤ 1;
* Having active central nervous system AML or AML of the APL/M3 subtype;
* History of keratitis;
* History of specified lung or renal disease;
* Having clinically significant cardiovascular disease;
* Known infection of Hepatitis B, C or E.

Key inclusion and exclusion criteria details are listed here, additional requirements may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2024-06-25 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities (dose escalation) | 21 days
Composite Complete Remission Rate (expansion) | Up to 24 months
  CR + CRh + CRi according ELN 2022 criteria

SECONDARY OUTCOMES:
Incidence and severity of adverse events | Up to 24 months
Number of patients with dose modifications | Up to 24 months
Rate of early death | Within 3 treatment cycles
Maximum Plasma Concentration (Cmax) BYON4413 | Up to 24 months
Time to Cmax (Tmax) BYON4413 | Up to 24 months
Area under the curve (AUC) BYON4413 | Up to 24 months
Percentage of patients with confirmed anti-BYON4413 antibodies | Up to 24 months
Composite Complete Remission Rate (dose escalation) | Up to 24 months
  CR + CRh + CRi according ELN 2022 criteria
Percentage of blasts in bone marrow change from baseline | Up to 24 months
Percentage of blasts in peripheral blood change from baseline | Up to 24 months
Objective response rate | Up to 24 months
  CR + CRh + CRi + MLFS + PR according ELN 2022 criteria
Duration of response | Up to 24 months
Relapse-free survival | Up to 24 months
Event-free survival | Up to 24 months
Time to response | Up to 24 months
Overall survival | Up to 24 months

CONTACTS AND LOCATIONS:
Locations (9):
- Belgium (2):
  - Het Ziekenhuisnetwerk Antwerpen, Antwerp
  - UZ Leuven, Leuven
- Universitair Medisch Centrum Groningen, Groningen, Netherlands
- Spain (6):
  - Institut Catala d'Oncologia, Badalona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital San Pedro de Alcantara, Cáceres
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario y Politecnico La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No